CLINICAL TRIAL: NCT02107898
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of Alirocumab in Heterozygous Familial Hypercholesterolemia or High Cardiovascular Risk Patients With Hypercholesterolemia Not Adequately Controlled With Their Lipid Modifying Therapy
Brief Title: Efficacy and Safety Evaluation of Alirocumab in Patients With Heterozygous Familial Hypercholesterolemia or High Cardiovascular Risk Patients With Hypercholesterolemia on Lipid Modifying Therapy (ODYSSEY JAPAN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC13672; U1111-1115-7486 (Other: UTN)
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Q2W (Placebo Comparator): Placebo (for alirocumab) every two weeks (Q2W) added to stable lipid-modifying therapy (LMT).
  Interventions: Drug: Placebo (for alirocumab); Drug: Lipid-Modifying Therapy (LMT)
- Alirocumab 75 mg/Up to 150 mg Q2W (Experimental): Alirocumab 75 mg Q2W added to stable LMT for 52 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when LDL-C levels above pre-specified threshold at Week 8 as defined in Japan Atherosclerosis Society (JAS) Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012 i.e.
  * ≥100 mg/dL (2.59 mmol/L) in heFH participants or in non-familial hypercholesterolemia (non-FH) participants who had a history of documented coronary heart disease (CHD)
  * ≥120 mg/dL (3.10 mmol/L) in non-FH participants who had a history of documented diseases or other risk factors as categorized in primary prevention category III
  Interventions: Drug: Alirocumab; Drug: Lipid-Modifying Therapy (LMT)

INTERVENTIONS:
Drug: Placebo (for alirocumab) — Solution for injection, one subcutaneous injection in the abdomen, thigh, or outer area of upper arm with an auto-injector.
  Arms: Placebo Q2W
Drug: Alirocumab — Solution for injection, one subcutaneous injection in the abdomen, thigh, or outer area of upper arm with an auto-injector.
  Other Names: SAR236553; REGN727; Praluent
  Arms: Alirocumab 75 mg/Up to 150 mg Q2W
Drug: Lipid-Modifying Therapy (LMT) — Statin (pravastatin, simvastatin, fluvastatin, atorvastatin, pitavastatin, rosuvastatin) at stable dose with or without other LMT as clinically indicated.

SUMMARY:
Primary Objective:

To demonstrate the reduction of low-density lipoprotein cholesterol (LDL-C) by alirocumab as add-on therapy to stable daily statin therapy with or without other lipid modifying therapy in comparison with placebo after 24 weeks of treatment in heterozygous familial hypercholesterolemia (HeFH) or high cardiovascular risk participants with hypercholesterolemia.

Secondary Objectives:

* To evaluate the effect of alirocumab in comparison with placebo on LDL-C after 12 weeks of treatment.
* To evaluate the effect of alirocumab on other lipid parameters.
* To evaluate the long-term effect of alirocumab in comparison with placebo on LDL-C after 52 weeks of treatment.
* To evaluate the safety and tolerability of alirocumab.
* To evaluate the development of anti-alirocumab antibodies.
* To evaluate the pharmacokinetics of alirocumab.

DETAILED DESCRIPTION:
Total duration per participant of approximately 63 weeks (14 months) (screening: 3 weeks, double-blind treatment period: 52 weeks, and follow-up period: 8 weeks).

ELIGIBILITY:
Inclusion criteria:

Participants with heterozygous familial hypercholesterolemia or non-familial hypercholesterolemia who were not adequately controlled with a stable daily dose of statin with or without other lipid modifying therapy, at stable dose prior to the screening visit (Week -3).

Exclusion criteria:

1. LDL-C <100 mg/dL (<2.59 mmol/L) at the screening visit in participants with heterozygous familial hypercholesterolemia or in participants with non-familial hypercholesterolemia who had a history of documented coronary heart disease as described in Japan Atherosclerosis Society (JAS) Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
2. LDL-C <120 mg/dL (<3.10 mmol/L) at the screening visit in participants with non-familial hypercholesterolemia who had a history of documented diseases or other risk factors as categorized in primary prevention category III as described in JAS Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
3. Not on a stable daily dose of lipid modifying therapy (including statin) within 4 weeks prior to the screening visit or between screening and randomization visits.
4. Age <20 years at the screening visit.

The above information is not intended to contain all considerations relevant to a participants' potential participation in a clinical trial.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (32):
- Japan (32):
  - Investigational Site Number 392016, Adachi-Ku
  - Investigational Site Number 392029, Adachi-Ku
  - Investigational Site Number 392024, Aki-Gun
  - Investigational Site Number 392012, Chūōku
  - Investigational Site Number 392013, Chūōku
  - Investigational Site Number 392032, Fukui-shi
  - Investigational Site Number 392004, Hakusan-Shi
  - Investigational Site Number 392028, Kaga-Shi
  - Investigational Site Number 392002, Kanazawa
  - Investigational Site Number 392005, Kanazawa
  - Investigational Site Number 392023, Kawanishi-Shi
  - Investigational Site Number 392009, Kisarazu-Shi
  - Investigational Site Number 392026, Kitakyushu-Shi
  - Investigational Site Number 392003, Komatsu-Shi
  - Investigational Site Number 392011, Kuki-Shi
  - Investigational Site Number 392017, Matsumoto-Shi
  - Investigational Site Number 392007, Mito
  - Investigational Site Number 392006, Moriya-Shi
  - Investigational Site Number 392018, Nagoya
  - Investigational Site Number 392014, Oota-Ku
  - Investigational Site Number 392019, Osaka
  - Investigational Site Number 392020, Osaka
  - Investigational Site Number 392022, Osaka
  - Investigational Site Number 392030, Osaka
  - Investigational Site Number 392027, Oyabe-Shi
  - Investigational Site Number 392010, Saitama-Shi
  - Investigational Site Number 392015, Shinjuku-Ku
  - Investigational Site Number 392031, Shizuoka
  - Investigational Site Number 392021, Suita-Shi
  - Investigational Site Number 392025, Takamatsu
  - Investigational Site Number 392008, Tsuchiura-Shi
  - Investigational Site Number 392001, Yamagata

REFERENCES:
- [Result] Teramoto T, Kobayashi M, Tasaki H, Yagyu H, Higashikata T, Takagi Y, Uno K, Baccara-Dinet MT, Nohara A. Efficacy and Safety of Alirocumab in Japanese Patients With Heterozygous Familial Hypercholesterolemia or at High Cardiovascular Risk With Hypercholesterolemia Not Adequately Controlled With Statins - ODYSSEY JAPAN Randomized Controlled Trial. Circ J. 2016 Aug 25;80(9):1980-7. doi: 10.1253/circj.CJ-16-0387. Epub 2016 Jul 22. PMID 27452202
- [Derived] Schmidt AF, Carter JL, Pearce LS, Wilkins JT, Overington JP, Hingorani AD, Casas JP. PCSK9 monoclonal antibodies for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD011748. doi: 10.1002/14651858.CD011748.pub3. PMID 33078867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 31 centers in Japan. A total of 319 participants were screened between March 2014 and July 2014, 103 of whom were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Randomization was stratified according to heterozygous familial hypercholesterolemia (heFH) population. Assignment to treatment arms was done using an Interactive Web Response System in 1:2 (Placebo: Alirocumab) ratio after confirmation of selection criteria. 216 participants were randomized.
Groups:
- Placebo Q2W: Placebo (for alirocumab) subcutaneous (SC) injection every two weeks (Q2W) added to stable lipid-modifying therapy (LMT) for 52 weeks.
- Alirocumab 75 mg/Up to 150 mg Q2W: Alirocumab 75 mg SC injection Q2W added to stable LMT for 52 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when low-density lipoprotein cholesterol (LDL-C) levels ≥ 100 mg/dL (2.59 mmol/L) or ≥ 120 mg/dL (3.10 mmol/L) at Week 8 according to Japan Atherosclerosis Society (JAS) Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
Period: Overall Study
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Started | 72 (Randomized) | 144 (Randomized)
Treated | 72 | 143
Completed | 66 | 132
Not Completed | 6 | 12
Not completed — Adverse Event | 4 | 7
Not completed — Poor compliance to protocol | 0 | 1
Not completed — Participant moved | 0 | 2
Not completed — Consent withdrawn by participant | 2 | 1
Not completed — Randomized but not treated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Q2W: Placebo (for alirocumab) SC injection Q2W added to stable LMT for 52 weeks.
- Alirocumab 75 mg/Up to 150 mg Q2W: Alirocumab 75 mg SC injection Q2W added to stable LMT for 52 weeks. Alirocumab dose up-titrated to 150 mg from Week 12 when LDL-C levels ≥ 100 mg/dL (2.59 mmol/L) or ≥ 120 mg/dL (3.10 mmol/L) at Week 8 according to JAS Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W | Total
Number analyzed (Participants) | 72 | 144 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.0) | 60.3 (9.7) | 60.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 60 | 85
  Male | 47 | 84 | 131
Calculated LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Calculated LDL-C in mg/dL from Friedewald formula (LDL-C = Total cholesterol - High-density lipoprotein cholesterol [HDL-C] - [Triglyceride/5]).
  mg/dL | 141.6 (26.7) | 140.9 (26.8) | 141.2 (26.7)
Calculated LDL-C in mmol/L [Mean (Standard Deviation); unit: mmol/L] | 3.668 (0.691) | 3.650 (0.693) | 3.656 (0.691)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - Intent-to-Treat (ITT Analysis)
Description: Adjusted least-squares (LS) means and standard errors at Week 24 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 24
Population: ITT population: all randomized participants with one baseline and at least one post-baseline calculated LDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 72 | 143
percent change | 1.6 (1.8) | -62.5 (1.3)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; Alirocumab group was compared to placebo group using an appropriate contrast statement; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -64.1, 95% CI 2-sided [-68.5 to -59.8] — Alirocumab vs. Placebo

2. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection) (on-treatment analysis).
Time Frame: From Baseline to Week 24
Population: Modified ITT (mITT) population: all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 71 | 143
percent change | 1.7 (1.7) | -63.7 (1.2)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.05 level; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -65.3, 95% CI 2-sided [-69.4 to -61.3] — Alirocumab vs. Placebo

3. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 72 | 143
percent change | -2.7 (1.6) | -64.2 (1.1)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -61.5, 95% CI 2-sided [-65.3 to -57.7] — Alirocumab vs. Placebo

4. Secondary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On-treatment Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 24
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 71 | 143
percent change | -2.8 (1.5) | -64.8 (1.1)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -62.1, 95% CI 2-sided [-65.8 to -58.3] — Alirocumab vs. Placebo

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B at Week 24 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo B value on- or off-treatment (Apo B ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 71 | 141
percent change | -1.6 (1.7) | -55.0 (1.2)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -53.3, 95% CI 2-sided [-57.5 to -49.1] — Alirocumab vs. Placebo

6. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 24
Population: Participants of the mITT population with one baseline and at least one post-baseline Apo-B value on-treatment (Apo B mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 70 | 140
percent change | -2.1 (1.7) | -55.9 (1.2)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -53.8, 95% CI 2-sided [-57.8 to -49.8] — Alirocumab vs. Placebo

7. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment (non-HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 72 | 143
percent change | 2.6 (1.6) | -54.9 (1.2)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -57.5, 95% CI 2-sided [-61.5 to -53.5] — Alirocumab vs. Placebo

8. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 24
Population: Participants of the mITT population with one baseline and at least one post-baseline non-HDL-C value on-treatment (non-HDL-C mITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 71 | 143
percent change | 2.6 (1.6) | -56.0 (1.1)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -58.6, 95% CI 2-sided [-62.3 to -54.8] — Alirocumab vs. Placebo

9. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline Total-C value on- or off-treatment (Total-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 72 | 143
percent change | 2.0 (1.3) | -39.5 (0.9)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -41.5, 95% CI 2-sided [-44.6 to -38.4] — Alirocumab vs. Placebo

10. Secondary Outcome: Percent Change From Baseline in Apo B at Week 12 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Apo B ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 71 | 141
percent change | -3.3 (1.5) | -54.6 (1.1)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -51.2, 95% CI 2-sided [-54.9 to -47.6] — Alirocumab vs. Placebo

11. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 24
Population: Non-HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 72 | 143
percent change | -1.7 (1.4) | -56.3 (1.0)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -54.5, 95% CI 2-sided [-57.9 to -51.1] — Alirocumab vs. Placebo

12. Secondary Outcome: Percent Change From Baseline in Total-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 24
Population: Total-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 72 | 143
percent change | -2.1 (1.1) | -41.1 (0.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = -39.0, 95% CI 2-sided [-41.7 to -36.4] — Alirocumab vs. Placebo

13. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C Goal at Week 24 - ITT Analysis
Description: Calculated LDL-C goal was defined as:
  * <100 mg/dL (2.59 mmol/L) for heFH or non-FH participants who had a history of documented congestive heart disease (CHD), or
  * <120 mg/dL (3.10 mmol/L) for non-FH participants who had a history of documented diseases (ischemic stroke, peripheral artery disease, chronic kidney disease or diabetes) or other risk factors as defined in JAS Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2012.
  Adjusted percentages at Week 24 were obtained from multiple imputation approach model for handling of missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on- or off-treatment were included in imputation model.
Time Frame: Up to Week 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 72 | 143
percentage of participants | 10.2 | 96.7
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 552.1, 95% CI 2-sided [105.6 to 2886.8] — Alirocumab vs. Placebo

14. Secondary Outcome: Percentage of Participants Reaching Calculated LDL-C Goal at Week 24 - On-Treatment Analysis
Description: Adjusted percentages at Week 24 were from multiple imputation approach model including available post-baseline on-treatment data from Week 4 to Week 24 (i.e. up to 21 days after last injection).
Time Frame: Up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 71 | 143
percentage of participants | 10.6 | 97.9
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Threshold for significance ≤ 0.05; Multiple imputation approach followed by logistic regression model; Odds Ratio (OR) = 1367.8, 95% CI 2-sided [137.8 to 13578.3] — Alirocumab vs. Placebo

15. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from a multiple imputation approach followed by robust regression model for handling of missing data. All available post-baseline data from Week 4 to Week 24 regardless of status on-or off-treatment were included in the imputation model.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 72 | 143
percent change | 2.5 (2.5) | -39.5 (1.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by a robust regression model; Adjusted Mean Difference = -42.0, 95% CI 2-sided [-48.0 to -36.0] — Alirocumab vs. Placebo

16. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24 - ITT Analysis
Description: Adjusted means and standard errors at Week 24 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 24 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 72 | 143
percent change | 6.7 (3.7) | -15.3 (2.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by a robust regression model; Adjusted Mean Difference = -22.0, 95% CI 2-sided [-30.9 to -13.1] — Alirocumab vs. Placebo

17. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment (HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 72 | 143
percent change | 2.1 (1.5) | 7.9 (1.1)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 5.8, 95% CI 2-sided [2.1 to 9.4] — Alirocumab vs. Placebo

18. Secondary Outcome: Percent Change From Baseline in Apo A1 at Week 24 - ITT Analysis
Description: as for outcome 5
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo A1 value on- or off-treatment (Apo A1 ITT population).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 71 | 141
percent change | -2.6 (1.6) | 1.4 (1.1)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0382, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 4.0, 95% CI 2-sided [0.2 to 7.9] — Alirocumab vs. Placebo

19. Secondary Outcome: Percent Change From Baseline in Lipoprotein (a) at Week 12 - ITT Analysis
Description: Adjusted means and standard errors at Week 12 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 4 to Week 24 regardless of status on-or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 72 | 143
percent change | -0.5 (2.4) | -41.9 (1.7)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by a robust regression model; Adjusted Mean Difference = -41.4, 95% CI 2-sided [-47.0 to -35.7] — Alirocumab vs. Placebo

20. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 12 - ITT Analysis
Description: as for outcome 19
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 72 | 143
percent change | 2.4 (3.7) | -13.1 (2.6)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0007, Regression, Robust — Threshold for significance ≤ 0.05; Multiple imputation approach followed by a robust regression model; Adjusted Mean Difference = -15.5, 95% CI 2-sided [-24.4 to -6.6] — Alirocumab vs. Placebo

21. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 24
Population: HDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 72 | 143
percent change | -1.8 (1.2) | 4.7 (0.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 6.5, 95% CI 2-sided [3.7 to 9.3] — Alirocumab vs. Placebo

22. Secondary Outcome: Percent Change From Baseline in Apo A1 at Week 12 - ITT Analysis
Description: as for outcome 10
Time Frame: From Baseline to Week 24
Population: Apo A1 ITT population.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 71 | 141
percent change | -4.8 (1.1) | 1.5 (0.8)
Statistical Analysis 1: Comparison: Placebo Q2W vs Alirocumab 75 mg/Up to 150 mg Q2W; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance ≤ 0.05; LS Mean Difference = 6.3, 95% CI 2-sided [3.6 to 9.0] — Alirocumab vs. Placebo

23. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 52 - ITT Analysis
Description: Adjusted LS means and standard errors at Week 52 from MMRM model including available post-baseline data from Week 4 to Week 52 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 52
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 72 | 143
Percent change | -3.6 (1.9) | -62.5 (1.4)

24. Other Pre Specified Outcome: Percent Change From Baseline in Calculated LDL-C at Week 52 - On-Treatment Analysis
Description: Adjusted LS means and standard errors at Week 52 were obtained from MMRM model including available post-baseline on-treatment data from Week 4 to Week 52 (i.e. up to 21 days after last injection).
Time Frame: From Baseline to Week 52
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo Q2W | Alirocumab 75 mg/Up to 150 mg Q2W
Number analyzed (Participants) | 71 | 143
Percent change | -3.4 (1.7) | -64.6 (1.2)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 60 post-treatment follow-up visit) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'treatment-emergent period' (the time from the first dose of study drug up to the last dose of study drug +70 days). Analysis was done on safety population that included randomized participants who actually received at least 1 dose or part of a dose of double-blind investigational medicinal product (IMP) injection.
Groups:
- Placebo Q2W: Participants exposed to placebo (for alirocumab) SC injection Q2W added to stable LMT (mean exposition of 50 weeks).
- Alirocumab 75 mg/ Up to 150 mg Q2W: Participants exposed to alirocumab 75 mg /up to 150 mg SC injection Q2W added to stable LMT (mean exposition of 50 weeks).
Arm/Group | Placebo Q2W | Alirocumab 75 mg/ Up to 150 mg Q2W
Serious Adverse Events (participants affected / at risk) | 9/72 | 10/143
Other Adverse Events (participants affected / at risk) | 44/72 | 97/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=72) | Alirocumab 75 mg/ Up to 150 mg Q2W (N=143)
Cellulitis (Infections and infestations) | 0 | 1
Muscle abscess (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 1
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Medical device discomfort (General disorders) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 2 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=72) | Alirocumab 75 mg/ Up to 150 mg Q2W (N=143)
Nasopharyngitis (Infections and infestations) | 26 | 65
Pharyngitis (Infections and infestations) | 4 | 9
Influenza (Infections and infestations) | 6 | 1
Seasonal allergy (Immune system disorders) | 5 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 12
Hypertension (Vascular disorders) | 5 | 9
Dental caries (Gastrointestinal disorders) | 1 | 9
Abdominal pain upper (Gastrointestinal disorders) | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 | 1
Injection site reaction (General disorders) | 3 | 18
Fall (Injury, poisoning and procedural complications) | 5 | 11
Contusion (Injury, poisoning and procedural complications) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.